CLINICAL TRIAL: NCT03211130
Title: Randomized Controlled Pilot Study of a SystemCHANGE™ Medication Adherence Intervention in Older Adult Stroke Survivors
Brief Title: Using SystemCHANGE™ to Enhance Medication Adherence in Older Adult Stroke Survivors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: Saint Luke's Health System (Other)
Responsible Party: Principal Investigator, Cynthia Russell, Professor, School of Nursing, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dissertation
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Stroke, Ischemic
Keywords: medication adherence; self-management; antithrombotic
MeSH Terms: conditions — Ischemic Stroke; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SystemCHANGE™ (Experimental)
  Interventions: Behavioral: SystemCHANGE™
- Attention-Control (Active Comparator)
  Interventions: Behavioral: Attention-Control

INTERVENTIONS:
Behavioral: SystemCHANGE™ — During the intervention phase, the PI will visit both groups of participants at home at baseline and telephone them three times (day 3 ±2 days and months 1 and 2). Refer to tables 1 and 2 for intervention details. Treatment participants will implement SystemCHANGE™ activities related to medication taking with the assistance of the PI while attention-control participants will receive patient education materials on stroke. Perceived health data will be collected during the intervention phase. A 1-month maintenance phase follows the intervention phase. Electronic medication monitoring continues, but no intervention is delivered to either group.
  Arms: SystemCHANGE™
Behavioral: Attention-Control — An experienced stroke nurse will deliver the attention control intervention. Table 3.2 shows the 2-month attention-control intervention. The stroke materials were developed by the Saint Luke's Marion Bloch Neuroscience Institute and are given to every stroke patient prior to dismissal. The PI will call participants at day 3 ±2 days, and months 1 and 2 to review chapter(s) from the book and answer questions about it. Interval, frequency, and setting are all exactly the same for the intervention and control groups. If the control participant raises questions about medications or medication-taking, PI will refer them to their Neurologist.
  Arms: Attention-Control

SUMMARY:
This study evaluated the feasibility and acceptability of using a SystemCHANGE intervention in older adult stroke survivors to improve medication adherence. Half the participants will receive the SystemCHANGE intervention, while the other half will receive the attention-control education intervention.

ELIGIBILITY:
Inclusion Criteria:

* age ≥50 years old
* receives post-stroke care with Saint Luke's Neurological Consultants
* prescribed at least 1, once a day, antithrombotic medication
* able to provide informed consent
* able to open an electronic cap
* able to self-administer medications
* has or has access to a telephone
* has no cognitive impairment as determined by a score of 4 or greater on The Six- item Screener (SIS).

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility | one point in time at the end of the maintenance phase which is 3 months after randomization into groups
  Open ended questionnaire

SECONDARY OUTCOMES:
Social Support | One day at beginning of Intervention phase. Once 1 day at beginning of Maintenance phase.
  The Social Support Appraisals Index (SS-A) is a 23-item self-administered, a self-report scale measuring the degree to which a person feels cared for, respected, and involved with family and friends. The scale had good reliability and validity (Cronbach α coefficients .90, .81, and .84) (Vaux et al., 1986).
Perceived Health | One day at beginning of Intervention phase. Once 1 day at beginning of Maintenance phase.
  Perceived health status will be measured by one question, "How is your health in general?" Participant select excellent, very good, good, fair, poor, or very poor. Perceived health status reflects people's overall perception of their health, including both physical and psychological dimensions.
Personal Systems Behaviors | One day at beginning of Intervention phase. Once 1 day at beginning of Maintenance phase.
  The Systems Thinking Survey (adapted for patients), a 20-item, 5-point Likert response scale measuring perceptions of personal system behaviors.
Medication Adherence | after randomization through end of maintenance phase for a total of 3 months
  MA data will be retrieved from the MEMS®cap which is a medication cap containing a battery and microelectronics that records the date and the time of each cap removal to create a medication "event" ("MEMS® Cap versatile adherence monitoring cap," n.d.).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L. Wessol, BSN, Principal Investigator — University of Missouri, Kansas City; Cynthia L. Russell, Ph.D., Study Chair — Professor
Locations (1):
- Jennifer Wessol, Parkville, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided